CLINICAL TRIAL: NCT02937714
Title: Effectiveness of School Based Intervention for Promoting Mental Health Literacy Among Teachers: A Randomized Controlled Trial
Brief Title: Effectiveness of School Based Intervention for Promoting Mental Health Literacy Among Teachers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KingEdwardMU
Record Dates: First submitted 2016-10-13; First posted 2016-10-19 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: School Mental Health Training of Teachers
Keywords: Teachers; mental health literacy; school mental health promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School mental health training (Experimental): Teachers Training workshop Workshop based on local adaptation of WHO-EMRO school mental health manual will be conducted in school. The duration of the workshop will be 3 days. Teachers can decline to participate or withdraw at any stage.
  Interventions: Other: School Mental Health training
- Wait list control group (No Intervention): Wait list control group of teachers in same schools. Half of teachers in the same school will be the wait list control group.

INTERVENTIONS:
Other: School Mental Health training — School based intervention (Teacher training intervention) is the teachers training program based on World Health Organization, Eastern Mediterranean Region (WHO-EMRO) School mental health manual draft (December 2014). Topics to be covered in training workshop include normal childhood development, behaviour management strategies for schools, life skills training, essential components for healthy schools, recognizing warning signs for common psychiatric and developmental disorders common to children and adolescents & school based interventions for various psychiatric problems
  Other Names: WHO-EMRO School Mental Health Manual Based Training
  Arms: School mental health training

SUMMARY:
Significantly higher prevalence of emotional and behavioural problems have been reported from Pakistan.This higher prevalence along with stigma of psychiatric problems and limited child & adolescent mental health services in Pakistan means that it is important to consider alternate methods for promoting psychological and emotional well-being of our youth. Schools can thus act as a natural platform for mental health promotion as schools context has almost as much impact on students' emotional health as the family context.

Teachers' role in the school mental health initiatives cannot be overemphasized. Teachers own knowledge and beliefs regarding mental health influence the way they respond to students mental health crisis. Recognizing the need for wider implementation of evidence based school mental health interventions in the region and to help in addressing the mental health literacy of educators in resource constrained settings, World Health Organization, Eastern Mediterranean Region (WHO-EMRO) has developed a concise and practical manual of school mental health in December 2014. In the absence of any "whole school approach" study from Pakistan focusing on teachers training and addressing all the various evidence based components of promotion of positive mental health, Investigators aim to conduct a pilot randomized controlled trial to assess effectiveness of training based on WHO-EMRO manual, in addition to its feasibility & acceptability in improving teachers' mental health literacy and self-efficacy in dealing with students mental health issues.

HYPOTHESIS:

For teachers:

* School mental health training intervention will significantly improve teacher's mental health literacy & self-efficacy compared to wait list control group.
* At 3 months follow-up, control group teachers' mental health literacy will also improve compared to baseline due to contamination of information provided, across groups within the same school.

All hypothesis pertains to individual level.

For students:

Mental health training of teachers would lead to an overall improvement in student's outcome measure (student's emotional and behavioural difficulties) at 3 months follow-up.

DETAILED DESCRIPTION:
Pakistan is the 6th most populous country of the world with population over 188 million; Almost 35% of population is under the age of 14. Country cannot afford to ignore mental health of this large group. School experiences are important for children emotional, psychological and social development World Health Organization (WHO) also identifies promotion of emotional health and well- being as a core feature of their Health promoting school initiative. Schools can play an important role in promoting positive mental health, reducing stigma, raising awareness among teachers, parents and children about mental health issues as well as identifying and supporting youth experiencing mental health difficulties. Furthermore, mental health initiatives in schools help teachers to feel less stressed and be more satisfied with their role and save costs. Educational interventions involving teachers have shown significant improvement in teachers knowledge and attitudes regarding mental health & better accuracy of teacher identification of children and adolescents with mental health problems. Although importance of schools for mental health promotion and early identification for mental health problems has been evident for quite some time, it is almost nonexistent in developing countries including Pakistan with only a handful of studies focusing one aspect of health promoting school or on one disorder. World Health Organization, Eastern Mediterranean Region (WHO-EMRO) has developed a concise and practical manual of school mental health in December 2014.This manual is primarily intended for all stakeholders involved in the educational process including teachers. It aims for helping educators to take practical steps that can be implemented at low costs in school settings.

OBJECTIVE:

To assess the effectiveness of locally adapted WHO school mental health Manual based intervention in improving mental health literacy among school teachers through a randomized controlled trial.

Secondary objectives include

1. To assess whether school mental health Manual based intervention leads to better self- efficacy among school teachers.
2. To determine if mental health training of teachers would lead to an indirect improvement in students outcome measure (emotional and behavioural difficulties) and school psychosocial environment.

STUDY PHASE 1: Interaction with key stakeholders to do a current situational analysis / identify priority problems.by using WHO Questionnaires & in depth Interviews.

STUDY PHASE 2: Randomized controlled trial to assess effectiveness, feasibility & acceptability of the adapted manual delivery in school settings.

STUDY PHASE 3: Process Evaluation by feedback from Teachers.

ELIGIBILITY:
Inclusion Criteria:

* All the teachers in the participating schools.
* Teachers of Grade 1-10 will be approached.
* Both Genders.

Exclusion Criteria:

* Lack of informed consent.
* Teachers who are leaving/ not planning to be in the school in 3 months' time.
* Teachers who have not been involved in active teaching in last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Teachers' knowledge | At the end of 3 days workshop
  Mental health literacy refers to a person's knowledge and beliefs about mental disorders, which in turn increases their ability to recognize, manage, or prevent the development or exacerbation of mental health problems. It has various elements including: 1) enhancing capacity to obtain and maintain good mental health; 2) enhancing understanding of mental disorders and their treatments; 3) decreasing stigma related to mental illness; 4) enhancing help-seeking efficacy. It will be assessed in the study using a self-administered questionnaire based on literature review and addressing various mental health literacy elements. Although main outcome time frame is post workshop but it will be reevaluated at 3 months time to see if change from baseline is seen.

SECONDARY OUTCOMES:
Teachers' Sense of Self Efficacy | At the end of 3 days workshop
  Teachers sense of efficacy scale(TSES) measures teachers assessment of their self-efficacy for teaching tasks as well as their other responsibilities. Efficacy in Student Engagement & Efficacy in Classroom Management subscales will be used to assess self efficacy of teachers. There are 8 statements & each statement is rated on 9 point Likert scale. It will also be reassessed at 3 months after the training workshop to assess if change from baseline is seen.
Students behavioural and emotional Problems | 3 months after the teachers training
  Self- reported Strengths and Difficulties questionnaire{SDQ} (11-16 years) will be used to assess students behavioural and emotional problems. SDQ measures 25 attributes, which are grouped in subscales of five items each, generating scores for conduct, hyperactivity, emotional, peer problems and prosocial behaviour. Statements are rated on a three point likert scale:0(not tue), 1(somewhat true) and 2(certainly true). All scales excluding the last are added to generate a total difficulties score (0-40). Total difficulties and categories scores can be coded in normal, borderline and abnormal categories.

OTHER OUTCOMES:
The School psycho-Social Profile | 3 months after the teachers training
  The School psycho-Social Profile Questionnaire (PSE ; WHO tools)will be completed by principals before and 3 months after the teacher training.

CONTACTS AND LOCATIONS:
Overall Officials: Nazish Imran, MRCPsych, Principal Investigator — King Edward Medical University
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Syed EU, Hussein SA, Mahmud S. Screening for emotional and behavioural problems amongst 5-11-year-old school children in Karachi, Pakistan. Soc Psychiatry Psychiatr Epidemiol. 2007 May;42(5):421-7. doi: 10.1007/s00127-007-0188-x. Epub 2007 Apr 21. PMID 17450455
- [Background] Weist, MD & Murray M. Advancing school mental health promotion globally. Advances in School Mental Health Promotion 2007; 1(1): 2-12.
- [Background] Durlak JA, Weissberg RP, Dymnicki AB, Taylor RD, Schellinger KB. The impact of enhancing students' social and emotional learning: a meta-analysis of school-based universal interventions. Child Dev. 2011 Jan-Feb;82(1):405-32. doi: 10.1111/j.1467-8624.2010.01564.x. PMID 21291449
- [Background] Skre I, Friborg O, Breivik C, Johnsen LI, Arnesen Y, Wang CE. A school intervention for mental health literacy in adolescents: effects of a non-randomized cluster controlled trial. BMC Public Health. 2013 Sep 23;13:873. doi: 10.1186/1471-2458-13-873. PMID 24053381
- [Background] Kutcher S, Wei Y, McLuckie A, Bullock L. Educator mental health literacy: a programme evaluation of the teacher training education on the mental health & high school curriculum guide. Advances in School Mental Health Promotion 2013;6(2):83-93 DOI: 10.1080/1754730X.2013.784615
- [Background] Rahman A, Mubbashar MH, Gater R, Goldberg D. Randomised trial of impact of school mental-health programme in rural Rawalpindi, Pakistan. Lancet. 1998 Sep 26;352(9133):1022-5. doi: 10.1016/s0140-6736(98)02381-2. PMID 9759745
- [Background] Syed EU, Hussein SA. Increase in teachers' knowledge about ADHD after a week-long training program: a pilot study. J Atten Disord. 2010 Jan;13(4):420-3. doi: 10.1177/1087054708329972. PMID 19474460
- [Derived] Imran N, Rahman A, Chaudhry N, Asif A. Effectiveness of a school-based mental health intervention for school teachers in urban Pakistan: a randomized controlled trial. Child Adolesc Psychiatry Ment Health. 2022 May 3;16(1):33. doi: 10.1186/s13034-022-00470-1. PMID 35505362
- [Derived] Imran N, Rahman A, Chaudhry N, Asif A. World Health Organization "School Mental Health Manual"-based training for school teachers in Urban Lahore, Pakistan: study protocol for a randomized controlled trial. Trials. 2018 May 24;19(1):290. doi: 10.1186/s13063-018-2679-3. PMID 29793553